CLINICAL TRIAL: NCT06491706
Title: The Association of Biological Sex and Long-term Outcomes in Older Patients With Physical Restraint at the Emergency Department
Brief Title: Long-term Outcomes in Older Patients With Physical Restraint
Status: Completed | Type: Observational
Sponsor: Beaujon Hospital (Other)
Responsible Party: Principal Investigator, Prabakar VAITTINADA AYAR, Principal Investigator, Beaujon Hospital
Other Study IDs: urgBjNpr
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-07

CONDITIONS: Physical Restraint; Gender Bias; Morality
Keywords: physical restraint; emergency department; biological sex; long-term mortality
MeSH Terms: conditions — Sexism; Emergencies; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: the was no intervention — there was no intervention in this observational study

SUMMARY:
The worldwide population is ageing. Biological sex is first and foremost a genetic modifier of disease. To prevent self-arm many techniques can be used in older patients. Among them coercive measure consisting of physical restraint (PR) is one of the techniques.

This study aims to assess the effects of the biological sex on the long-term survival after PR in geriatric patients during the initial emergency department (ED) visit.

This retrospective study included patients between November 2019 to March 2021. All consecutive hospitalized patients after emergency department visit older than 75 years with PR were included.

The population was compared according to the biological sex. One-year all-cause mortality was plotted with the Kaplan-Meier curve. Hazard ratios (HRs) for 1-year mortality were calculated using a Cox proportional hazards regression model. Mortality was monitored over a 3-year period.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive older patients ≥ 75-year-old hospitalized to the observation unit or to the ward from the ED
* If physical restraint were mentioned in medical records

Exclusion Criteria:

* if patients were less than 75 years old
* Without physical restraint
* Not hospitalized
* If a patient was admitted more than once, only the first episode was taken as index admission

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Study Population: All consecutive older patients ≥ 75-year-old
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
one year mortaliy | ONE year

CONTACTS AND LOCATIONS:
Overall Officials: Prabakar VAITTINADA AYAR, MD, PhD, Principal Investigator — Hôpital Beaujon
Locations (1):
- Hopital BEAUJON, Clichy, France

IPD SHARING:
Plan to Share IPD: Yes